CLINICAL TRIAL: NCT02669342
Title: Randomized Controlled Trial for the Early Clinical Experience and Evaluation of the Radiance Clear Sharklet Silicone Foley Catheter
Brief Title: Sharklet Catheter Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Dirk Lange, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H15-03435
Record Dates: First submitted 2016-01-20; First posted 2016-02-01 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Urinary Catheter; Urinary Tract Infections
Keywords: Infection; Urinary Catheter; Sharklet
MeSH Terms: conditions — Urinary Tract Infections; Infections

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients are not told which catheter is inserted at which time point until after they exit the study.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Sharklet Catheter for 2 weeks first (Active Comparator): Arm A will have catheters inserted according to the schedule below:
  1. Sharklet catheter inserted for 2 weeks
  2. Standard catheter inserted for 2 weeks
  3. Sharklet catheter inserted for 4 weeks
  4. Standard catheter inserted for 4 weeks
  Interventions: Device: Radiance™ Clear Sharklet® Silicone Foley Catheter; Device: Silicone Foley Catheter
- Group B: Sharklet Catheter for 4 weeks first (Active Comparator): Arm B will have catheters inserted according to the schedule below:
  1. Sharklet catheter inserted for 4 weeks
  2. Standard catheter inserted for 4 weeks
  3. Sharklet catheter inserted for 2 weeks
  4. Standard catheter inserted for 2 weeks
  Interventions: Device: Radiance™ Clear Sharklet® Silicone Foley Catheter; Device: Silicone Foley Catheter

INTERVENTIONS:
Device: Radiance™ Clear Sharklet® Silicone Foley Catheter
Device: Silicone Foley Catheter
  Other Names: Standard of care

SUMMARY:
The aim of this study is to determine if the Sharklet catheter, with its unique coating, reduces infections in participants, when compared to a standard catheter.

DETAILED DESCRIPTION:
The aim of this study is to determine if the Sharklet catheter, with its unique coating, reduces infections in participants, when compared to a standard catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires a chronic indwelling Foley catheter for at least 14 days. Catheters will not remain indwelling greater than 30 days at a time
* Patient is more than 19 years of age
* Patient is able to give informed consent
* Patient is able to attend follow-up sessions

Exclusion Criteria:

* Patient is less than 19 years of age
* Patient is pregnant
* Patient with a known allergy to silicone
* Patient has urinary tract anatomic abnormality that would prevent placement of a standard Foley catheter
* Patient unable to accommodate the catheter
* Patient has an active urinary tract infection (UTI) or other diagnosed infection that is untreated. Once the infection has been treated, the patient is eligible for study.
* Patient currently taking (or expected to take) more than a single dose of antibiotics for prevention of other infections during the catheter indwell period
* Patient has uncontrolled fecal incontinence (uncontrolled stool/poop passage)
* Patient is unable to feel and/or communicate their symptoms
* Informed consent is unable to be obtained
* Patient is unable or unwilling to comply with the study follow-up schedule
* Patient has a medical condition or disorder that would limit life expectancy to less than 30 days or that may cause non-compliance with the protocol or confound the data analysis
* Any other reason that if in the opinion of the investigator would make the patient unsuitable for enrollment in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Catheter scrapings examined for colonization/biofilm burden and compared to the urine screen collected from the participant (cfu/mL) | 12 weeks
  Determine if there will be less adherent bacteria/biofilm to the Sharklet catheter compared to the controls.
Number of symptomatic Urinary tract infections (UTIs) determined by urine culture | 12 weeks
  Determine number of symptomatic UTIs between the 2 groups as determined by urine culture.

SECONDARY OUTCOMES:
Delay to symptomatic CA-SUTI | 12 weeks
  Delay to symptomatic catheter-associated symptomatic urinary tract infection (CA-SUTI)
Incidence of bacteria | 12 weeks
  Incidence of bacteremia following CA-SUTI
Incidence of Crustation | 12 weeks
  Incidence of catheter obstruction/encrustation requiring removal
Incidence of Discomfort | 12 weeks
  Incidence of significant discomfort/pain requiring removal
Surface analysis of the type of bacteria found on each catheter | 12 weeks
  Surface analysis (e.g., SEM) of removed catheters for qualitative assessment of bacterial colonization
Surface analysis of the amount of encrustation | 12 weeks
  Surface analysis (e.g., SEM) of removed catheters for qualitative assessment of encrustation
Surface analysis of the biofilm formation | 12 weeks
  Surface analysis (e.g., SEM) of removed catheters for qualitative assessment of biofilm formation

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Lange, PhD, Principal Investigator — University of British Columbia
Locations (1):
- The Stone Centre, VGH/UBC, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No